CLINICAL TRIAL: NCT03282994
Title: Evaluation of the Dermal Cooling System for Cryotherapy of Common Skin Conditions
Brief Title: Dermal Cooling System for Cryotherapy of Common Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-17-003
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment with cryotherapy (Experimental): Dermal Cooling System
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Cryotherapy

SUMMARY:
Prospective, non-randomized, open-label study to evaluate the dermal cooling system for cryotherapy of common skin conditions.

DETAILED DESCRIPTION:
The purpose of this study is to establish that controlled localized cooling with the Dermal Cooling System will elicit an improvement in the cosmetic appearance of benign superficial lesions associated with common skin conditions that are currently being treated with cryosurgical methods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has benign superficial lesion(s) associated with common skin conditions amenable to cryosurgical treatment including, for example, psoriasis, acne, rosacea, and sebaceous hyperplasia.
3. Subject is willing to have up to 40 test sites treated.
4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Physician prescribed procedures in the area of intended treatment in the previous 6 months (e.g., photodynamic therapy, intense pulsed light therapy, laser surgery).
2. Dermatological conditions (e.g. vitiligo, open wounds, infection, pre-cancerous or malignant lesions) in the location of the treatment sites that would, in the professional opinion of the investigator, potentially pose an increased risk to the subject.
3. History of melanoma.
4. Known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease).
5. History of abnormal wound healing or abnormal scarring
6. Inability or unwillingness to comply with the study requirements.
7. Subject is pregnant or planning to become pregnant while enrolled in the study.
8. Subject is lactating.
9. Current enrollment in a clinical study of any other unapproved investigational drug or device.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an increased or unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
Improvement in appearance in the treatment area | 3-months
  Improvement in appearance in the treated area at the 3-month follow-up visit, as determined by the Physician Global Assessment (PGA).

SECONDARY OUTCOMES:
Incidence of procedure related adverse events | less than 12 months
  • Safety of the treatment as determined by the incidence of device- or procedure-related serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Tatsutani, PhD, Study Director — R2 Dermatology
Locations (3):
- United States (3):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Zel Skin and Laser Specialists, Edina, Minnesota
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No